CLINICAL TRIAL: NCT04566861
Title: Biological Processes Underlying Anxiety During Pregnancy: A Substudy of an Anxiety-focused Early Prenatal Intervention for the Prevention of Common Mental Disorders in Pakistan
Brief Title: Happy Mother - Healthy Baby: Supplement Study on Biological Processes Underlying Anxiety During Pregnancy
Acronym: HMHB-Bio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Human Development Research Foundation, Pakistan (Other); Rawalpindi Medical College, Pakistan (Other); University of Liverpool (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 3R01MH111859-03S1 (NIH); 3R01MH111859-03S1 (NIH)
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Anxiety
Keywords: randomized controlled trial; inflammation; hormones
MeSH Terms: conditions — Anxiety Disorders; Inflammation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Within women in a larger randomized trial (randomized to the intervention or enhanced care group), we propose to study biological correlates of antenatal anxiety (i.e., immune and endocrine functioning) in 300 women: in addition to 200 drawn from our randomized trial (100 intervention, 100 usual care), we will also include 100 healthy women without anxiety or depression. These enrollment goals were modified after interruptions by the Covid-19 pandemic.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigators and outcomes assessors will be blind to the randomization status of the 200 anxious women assigned to the intervention and enhanced usual care groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anxious pregnant women - intervention group (Experimental): 100 pregnant women who have at least mild anxiety will be randomized to the intervention group where they will receive six one-on-one core sessions of Cognitive Behavioral Therapy during pregnancy (plus possible booster sessions)
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT) for anxiety during pregnancy
- Anxious pregnant women - enhanced usual care group (No Intervention): 100 pregnant women who have at least mild anxiety will be randomized to the enhanced usual care group. Reminder calls were given, provider visits were facilitated (shorter wait times), and transportation to assist participants in attending appointments and medically indicated ultrasounds were paid for (as in the other group).
- Non-anxious pregnant women - healthy control (No Intervention): 100 pregnant women who do not have symptoms of anxiety or depression be followed in the healthy control group. Reminder calls were given, provider visits were facilitated (shorter wait times), and transportation to assist participants in attending appointments and medically indicated ultrasounds were paid for (as in the other groups).

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) for anxiety during pregnancy — Women who are randomized to the intervention group will receive six core Cognitive Behavioral Therapy (CBT) sessions for anxiety during pregnancy (and possible booster sessions) to treat symptoms of anxiety.
  Arms: Anxious pregnant women - intervention group

SUMMARY:
As a supplement to the ongoing randomized evaluation of the Cognitive Behavioral Therapy (CBT) anxiety prevention intervention in Pakistan (R01-MH111859), the investigators propose to explore potential biological mechanisms (related to inflammation and endocrine functioning) of antenatal anxiety through additional data collection with 300 pregnant women.

DETAILED DESCRIPTION:
This study will leverage the ongoing randomized evaluation of the CBT anxiety prevention intervention in Pakistan (R01-MH111859) to explore potential biological mechanisms. This CBT intervention targets both sub-threshold anxiety symptoms and generalized anxiety disorder (GAD) in early- to mid- pregnancy, aiming to both prevent and treat Common Mental Disorders (CMDs) (GAD and major depressive episodes (MDE)) as well as improve birth outcomes. The study team proposes to additionally study biological correlates of antenatal anxiety (i.e., immune and endocrine functioning) in 300 women: in addition to 200 drawn from our randomized trial (100 intervention, 100 usual care), the study will also include 100 healthy women without anxiety or depression. The aims are to 1) characterize the "immune phenotype" of anxious women across the peripartum, specifically by measuring the relation among anxiety symptoms and peripheral markers of inflammation within and across women (both anxious and healthy) and between those receiving the intervention and control; 2) determine the relation between levels of allopregnanolone (ALLO) in pregnancy and concurrent anxiety symptoms and future symptoms of postpartum depression (PPD), 3) examine the relation between changes in immune functioning and ALLO levels in anxious pregnancy across time, 4) examine whether immune function and/or ALLO are mediators or moderators of the association between antenatal anxiety and preterm birth and/or small-for-gestational age, and 5) examine the effects of both anxiety and the intervention (including biomarkers) on infant development at six weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* ability to understand spoken Urdu
* pregnant, ≤22 weeks' gestation
* age ≥18 years
* residence ≤20 km of Holy Family Hospital
* intent to reside in the study areas until the completion of the study

Exclusion Criteria:

* Current anemia
* Current major depressive episode (MDE on SCID) or life-threatening health conditions including e.g. active severe depression or suicidal ideation
* Self-report of past or current significant learning disability
* Self-report of past or current psychiatric disorder (e.g. bipolar disorder or schizophrenia) or psychiatric care (e.g. current use of anxiolytic drug and/or other psychotropic drug)
* medical disorders or severe maternal morbidity that require inpatient management that would preclude participation (101)
* ICU admission indicated by diagnosis (not only for assessment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women and their children
Enrollment: 117 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela J Surkan, ScD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Holy Family Hospital, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified project data from the study will be posted on ClinicalTrials.gov and the National Institute of Mental Health (NIMH) data archive.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol, statistical analysis plan and informed consent form are available upon request now.
Access Criteria: The can be access upon request from the study PI: psurkan@jhu.edu

REFERENCES:
- [Background] Atif N, Nazir H, Zafar S, Chaudhri R, Atiq M, Mullany LC, Rowther AA, Malik A, Surkan PJ, Rahman A. Development of a Psychological Intervention to Address Anxiety During Pregnancy in a Low-Income Country. Front Psychiatry. 2020 Jan 10;10:927. doi: 10.3389/fpsyt.2019.00927. eCollection 2019. PMID 31998151
- [Background] Sherer ML, Malik A, Osborne LM, Rowther AA, Zaidi A, Atif N, Rahman A, Kahloon LE, Salman M, Yenokyan G, Surkan PJ. Biological Mechanisms in Pregnant Women With Anxiety (Happy Mother-Healthy Baby Supplement Study): Protocol for a Longitudinal Mixed Methods Observational Study. JMIR Res Protoc. 2023 Apr 11;12:e43193. doi: 10.2196/43193. PMID 37040167
- [Result] Surkan PJ, Hamdani SU, Huma ZE, Nazir H, Atif N, Rowther AA, Chaudhri R, Zafar S, Mullany LC, Malik A, Rahman A. Cognitive-behavioral therapy-based intervention to treat symptoms of anxiety in pregnancy in a prenatal clinic using non-specialist providers in Pakistan: design of a randomised trial. BMJ Open. 2020 Apr 15;10(4):e037590. doi: 10.1136/bmjopen-2020-037590. PMID 32300002
- [Derived] Etyemez S, Mehta K, Tutino E, Zaidi A, Atif N, Rahman A, Malik A, Voegtline KM, Surkan PJ, Osborne LM. The immune phenotype of perinatal anxiety in an anxiety-focused behavioral intervention program in Pakistan. Brain Behav Immun. 2024 Aug;120:141-150. doi: 10.1016/j.bbi.2024.05.028. Epub 2024 May 21. PMID 38777289

RESULTS

PARTICIPANT FLOW:
Groups:
- Anxious Pregnant Women - Enhanced Usual Care Group: 100 pregnant women who have at least mild anxiety will be randomized to the enhanced usual care group. They will not receive intervention sessions but will receive transportation vouchers to come to the hospital and facilitation by study staff to attend to their regular antenatal care visits.
- Non-anxious Pregnant Women - Healthy Control: 100 pregnant women who do not have symptoms of anxiety or depression be followed in the healthy control group. They will not receive intervention sessions but will receive transportation vouchers to come to the hospital and facilitation by study staff to attend to their regular antenatal care visits.
Period: Overall Study
Arm/Group | Anxious Pregnant Women - Intervention Group | Anxious Pregnant Women - Enhanced Usual Care Group | Non-anxious Pregnant Women - Healthy Control
Started | 26 | 31 | 60
Completed | 17 | 19 | 42
Not Completed | 9 | 12 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anxious Pregnant Women - Intervention Group | Anxious Pregnant Women - Enhanced Usual Care Group | Non-anxious Pregnant Women - Healthy Control | Total
Number analyzed (Participants) | 26 | 31 | 60 | 117
Age, Continuous [Mean (Full Range); unit: Years] | 25.65 [18 to 37] | 24.74 [18 to 33] | 26.27 [20 to 38] | 25.73 [18 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 31 | 60 | 117
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 26 | 31 | 60 | 117
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Pakistan | 26 | 31 | 60 | 117
Baseline Hospital Anxiety&Depression Score (HADS) of >=8 on the anxiety subscale for anxious group [Number; unit: participants] | 26 | 31 | 0 | 57

OUTCOME MEASURES:

1. Primary Outcome: Peripheral Markers of Inflammation
Description: Differences in levels of peripheral inflammatory markers and change in these markers across time (trimester 1 (T1), trimester 2 (T2), trimester 3 (T3) and postpartum (PP)) between anxious and healthy women, and between intervention and control women. Markers include IFNgamma, IL6, IL8, IL10, IL12p70, TNFalpha, IL17A, TARC, MIP1alpha, MCP4, Eotaxin
Time Frame: trimester 1, trimester 2, trimester 3, 6 weeks postpartum
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Anxious Pregnant Women - Intervention Group | Anxious Pregnant Women - Enhanced Usual Care Group | Non-anxious Pregnant Women - Healthy Control
Number analyzed (Participants) | 26 | 31 | 60
pg/ml
  TARC at T1 | 17.09 (10.30) | 20.22 (10.85) | 14.79 (8.06)
  TARC at T2 | 11.78 (8.30) | 12.12 (7.18) | 11.65 (7.87)
  TARC at T3 | 6.06 (2.95) | 7.52 (3.29) | 6.65 (3.35)
  TARC at PP | 15.28 (6.40) | 18.07 (8.84) | 16.81 (11.03)
  MIP1alpha at T1 | 2.52 (1.61) | 2.17 (0.75) | 2.16 (0.74)
  MIP1alpha at T2 | 4.09 (4.33) | 2.93 (1.45) | 3.41 (1.43)
  MIP1alpha at T3 | 2.45 (0.99) | 2.22 (0.60) | 2.28 (1.02)
  MIP1alpha at PP | 3.62 (0.83) | 3.23 (0.83) | 3.54 (0.99)
  MCP4 at T1 | 45.70 (28.30) | 57.08 (33.28) | 42.32 (20.64)
  MCP4 at T2 | 35.46 (24.07) | 41.26 (20.78) | 33.27 (16.69)
  MCP4 at T3 | 25.89 (13.96) | 30.10 (14.83) | 22.86 (8.61)
  MCP4 at PP | 72.87 (27.65) | 67.84 (25.82) | 65.53 (29.78)
  Eotaxin at T1 | 157.87 (65.20) | 178.82 (75.27) | 140.11 (66.73)
  Eotaxin at T2 | 112.06 (46.94) | 141.96 (70.10) | 101.17 (39.15)
  Eotaxin at T3 | 58.00 (23.23) | 72.12 (25.54) | 55.80 (24.26)
  Eotaxin at PP | 222.59 (91.64) | 187.66 (78.50) | 182.52 (73.72)
  IL17A at T1 | 1.01 (1.26) | 1.28 (1.44) | 1.06 (1.14)
  IL17A at T2 | 1.15 (1.67) | 0.90 (0.85) | 0.81 (0.55)
  IL17A at T3 | 1.19 (1.29) | 1.12 (7.98) | 1.26 (3.05)
  IL17A at PP | 2.08 (2.29) | 1.56 (0.85) | 2.64 (4.67)
  IFN gamma at T1 | 8.85 (15.44) | 6.77 (7.98) | 5.27 (3.49)
  IFN gamma at T2 | 6.09 (4.07) | 7.57 (9.55) | 6.07 (3.98)
  IFN gamma at T3 | 4.67 (3.61) | 4.44 (2.34) | 4.53 (3.35)
  IFN gamma at PP | 14.64 (21.57) | 10.50 (9.13) | 8.27 (9.50)
  IL6 at T1 | 0.38 (0.13) | 0.39 (0.22) | 0.42 (0.19)
  IL6 at T2 | 0.44 (0.19) | 0.44 (0.40) | 0.48 (0.24)
  IL6 at T3 | 0.63 (0.27) | 0.55 (0.32) | 0.64 (0.48)
  IL6 at PP | 0.58 (0.21) | 0.59 (0.37) | 0.66 (0.36)
  IL8 at T1 | 1.94 (0.62) | 2.09 (1.04) | 1.89 (0.72)
  IL8 at T2 | 1.69 (0.67) | 2.12 (1.27) | 1.91 (0.81)
  IL8 at T3 | 2.09 (1.22) | 2.32 (0.91) | 2.03 (0.81)
  IL8 at PP | 3.28 (1.40) | 3.45 (0.92) | 3.33 (1.68)
  IL10 at T1 | 0.17 (0.10) | 0.23 (0.36) | 0.20 (0.13)
  IL10 at T2 | 0.16 (0.06) | 0.21 (0.14) | 0.26 (0.36)
  IL10 at T3 | 0.26 (0.20) | 0.19 (0.09) | 0.25 (0.31)
  IL10 at PP | 0.30 (0.35) | 0.22 (0.15) | 0.21 (0.20)
  IL12P70 at T1 | 0.04 (0.03) | 0.05 (0.03) | 0.51 (0.03)
  IL12P70 at T2 | 0.04 (0.03) | 0.05 (0.04) | 0.07 (0.04)
  IL12P70 at T3 | 0.05 (0.03) | 0.04 (0.04) | 0.05 (0.03)
  IL12P70 at PP | 0.05 (0.05) | 0.04 (0.06) | 0.06 (0.09)
  TNFalpha at T1 | 0.69 (0.14) | 0.65 (0.14) | 0.65 (0.16)
  TNFalpha at T2 | 0.74 (0.13) | 0.75 (0.25) | 0.81 (0.21)
  TNFalpha at T3 | 0.94 (0.23) | 0.86 (0.22) | 0.98 (0.33)
  TNFalpha at PP | 1.29 (0.44) | 1.11 (0.26) | 1.12 (0.27)

2. Primary Outcome: Allopregnanolone Levels and Anxiety Symptoms Across the Peripartum
Description: Measure differences in level of allopregnanolone (mean) at each time point and across time (trimester 1 (T1), trimester 2 (T2), trimester 3 (T3) and postpartum (PP)) between anxious women and healthy women, and between intervention and control.
  The results are measured by log-transformed values of the concentration of each cytokine in the plasma, in ng/mL (nanogram per milliliter).
Time Frame: trimester 2, trimester 3, 6 weeks postpartum
Population: trimester 2, trimester 3, 6 weeks postpartum
Measure: Mean (Standard Deviation); unit: log (ng/ml)
Arm/Group | Anxious Pregnant Women - Intervention Group | Anxious Pregnant Women - Enhanced Usual Care Group | Non-anxious Pregnant Women - Healthy Control
Number analyzed (Participants) | 21 | 25 | 50
log (ng/ml)
  Allopregnanolone at T2 | -0.3796214 (0.7621596) | -0.3828328 (0.8335611) | -0.2820709 (0.9410302)
  Allopregnanolone at T3 | 2.825177 (0.995552) | 3.149545 (0.3715666) | 3.048794 (0.3715666)
  Allopregnanolone at W6 | -0.592519 (0.5954829) | -0.6423627 (0.5764104) | -0.7948805 (0.4380674)

3. Primary Outcome: Allopregnanolone Levels Predicting Postpartum Depression
Description: Differences in allopregnanolone levels at the second trimester between women who do and do not go on to develop postpartum depression (PPD).
  The results are measured by log-transformed values of the concentration of allopregnanolone in the plasma, in ng/ml (nanogram per milliliter.
  Women who have Allopregnanolone (ALLO) levels and developed PPD are analyzed.
Time Frame: Trimester 2
Population: Trimester 2. The numbers of analyzed data is lower than the overall number since not every women who had ALLO had also data available for PPD.
Measure: Mean (Standard Deviation); unit: log (ng/ml)
Arm/Group | Anxious Pregnant Women - Intervention Group | Anxious Pregnant Women - Enhanced Usual Care Group | Non-anxious Pregnant Women - Healthy Control
Number analyzed (Participants) | 19 | 21 | 41
log (ng/ml)
  Allopregnanolone at T2 in women with PPD: number analyzed (Participants) | 4 | 8 | 0
  Allopregnanolone at T2 in women with PPD | -0.004127186 (0.7631303) | -0.8292861 (0.7694288) |
  Allopregnanolone at T2 in women without PPD: number analyzed (Participants) | 15 | 13 | 41
  Allopregnanolone at T2 in women without PPD | -0.4591347 (0.7616261) | -0.08843005 (0.7569726) | -0.1739193 (0.9115309)

4. Primary Outcome: Allopregnanolone (ALLO) and Immune Function
Description: Measure the relationship between ALLO levels and levels of peripheral inflammatory markers across time (trimester 2 (T2), trimester 3 (T3) and 6 weeks postpartum (W6))
Time Frame: trimester 2, trimester 3, 6 weeks postpartum
Population: Trimester 2, 3, postpartum
Measure: Number; unit: p value
Arm/Group | Anxious Pregnant Women - Intervention Group | Anxious Pregnant Women - Enhanced Usual Care Group | Non-anxious Pregnant Women - Healthy Control
Number analyzed (Participants) | 21 | 25 | 50
p value
  T2 Allo and T2_EOTAXIN | 0.607838873 | 0.508436643 | 0.731221724
  T2 Allo and T2_IFNgam | 0.943495625 | 0.962951805 | 0.32767424
  T2 Allo and T2_IL10 | 0.442764509 | 0.852343415 | 0.251810201
  T2 Allo and T2_IL12P70 | 0.043026211 | 0.182583506 | 0.032112919
  T2 Allo and T2_IL17A | 0.994071069 | 0.628278059 | 0.155033717
  T2 Allo and T2_IL6 | 0.661240061 | 0.433900134 | 0.101928485
  T2 Allo and T2_IL8 | 0.58507263 | 0.377422318 | 0.000902406
  T2 Allo and T2_MCP4 | 0.253876939 | 0.975614712 | 0.261553
  T2 Allo and T2_MIP1alp | 0.211464436 | 0.219395666 | 0.757648777
  T2 Allo and T2_TARC | 0.044208627 | 0.09877797 | 0.482216914
  T2 Allo and T2_TNFalp | 0.620118634 | 0.452187217 | 0.389716682
  T3 Allo and T3_EOTAXIN | 0.438406999 | 0.484822182 | 0.644129208
  T3 Allo and T3_IFNgam | 0.404728602 | 0.373945489 | 0.747287036
  T3 Allo and T3_IL10 | 0.119629591 | 0.335957072 | 0.299247829
  T3 Allo and T3_IL12P70 | 0.933378078 | 0.337344443 | 0.898094409
  T3 Allo and T3_IL17A | 0.771455608 | 0.280587079 | 0.412507598
  T3 Allo and T3_IL6 | 0.663796915 | 0.083926433 | 0.526805187
  T3 Allo and T3_IL8 | 0.681722947 | 0.570578156 | 0.447858
  T3 Allo and T3_MCP4 | 0.725048008 | 0.420134106 | 0.090351732
  T3 Allo and T3_MIP1alp | 0.40714722 | 0.241913557 | 0.454254606
  T3 Allo and T3_TARC | 0.12961388 | 0.420828347 | 0.604242922
  T3 Allo and T3_TNFalp | 0.25342432 | 0.921598373 | 0.981377152
  W6 Allo and W6_EOTAXIN | 0.056363143 | 0.488055787 | 0.00049734
  W6 Allo and W6_IFNgam | 0.778831242 | 0.493655855 | 0.019717559
  W6 Allo and W6_IL10 | 0.380554726 | 0.706511155 | 0.038619177
  W6 Allo and W6_IL12P70 | 0.434897804 | 0.707672478 | 0.086203475
  W6 Allo and W6_IL17A | 0.803123246 | 0.514072112 | 0.132466231
  W6 Allo and W6_IL6 | 0.653576209 | 0.999655946 | 0.174873815
  W6 Allo and W6_IL8 | 0.965403419 | 0.224965514 | 0.183430195
  W6 Allo and W6_MCP4 | 0.752085053 | 0.54436977 | 0.42633973
  W6 Allo and W6_MIP1alp | 0.134643876 | 0.277197163 | 0.571967334
  W6 Allo and W6_TARC | 0.065203743 | 0.923420368 | 0.922589566
  W6 Allo and W6_TNFalp | 0.286463458 | 0.694997299 | 0.965333979

5. Secondary Outcome: Birth Outcomes
Description: Differences in birth outcomes (preterm birth, small for gestational age, low birth weight) between women with high inflammatory markers vs. those low in inflammatory markers, and also between anxious and healthy women.
Time Frame: at birth
Population: The number analyzed is different than the overall number because data was not collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Anxious Pregnant Women - Intervention Group | Anxious Pregnant Women - Enhanced Usual Care Group | Non-anxious Pregnant Women - Healthy Control
Number analyzed (Participants) | 26 | 31 | 60
Participants
  preterm birth: number analyzed (Participants) | 20 | 20 | 25
  preterm birth | 5 | 3 | 3
  small for gestational age: number analyzed (Participants) | 20 | 20 | 25
  small for gestational age | 5 | 6 | 8
  low birth weight: number analyzed (Participants) | 23 | 23 | 49
  low birth weight | 11 | 8 | 13

6. Secondary Outcome: Infant Neuro-development Using Ages & Stages Questionnaire, Third Edition (ASQ-3)
Description: Measure infant neuro-development using Ages & Stages Questionnaire to measure differences in infant neurodevelopment (communication, gross motor, fine motor, personal-social and problem solving) using a standardized questionnaire between those high in inflammatory markers vs. those low, and also between anxious and healthy women
  communication cut-off score 22.77 gross motor cut-off score 41.84 fine motor cut-off score 30.16 personal-social cut-off score 24.62 problem solving cut-off score 33.71
  Number of participants with impaired neuron-developmental infants (below cut-off scores) are reported below
Time Frame: 6 weeks postpartum
Population: The number analyzed is different than the overall number because data was not collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Anxious Pregnant Women - Intervention Group | Anxious Pregnant Women - Enhanced Usual Care Group | Non-anxious Pregnant Women - Healthy Control
Number analyzed (Participants) | 26 | 31 | 60
Participants
  communication below cut-off score: number analyzed (Participants) | 20 | 20 | 24
  communication below cut-off score | 0 | 0 | 0
  gross motor below cut-off score | 3 | 2 | 1
  fine motor below cut-off score | 1 | 0 | 0
  personal-social below cut-off score | 1 | 0 | 0
  problem solving below cut-off score | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 months
Description: We only had still births, miscarriages and child deaths of the participants who were giving births
Arm/Group | Anxious Pregnant Women - Intervention Group | Anxious Pregnant Women - Enhanced Usual Care Group | Non-anxious Pregnant Women - Healthy Control
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/31 | 0/60
Serious Adverse Events (participants affected / at risk) | 9/26 | 14/31 | 20/60
Other Adverse Events (participants affected / at risk) | 0/26 | 0/31 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anxious Pregnant Women - Intervention Group (N=26) | Anxious Pregnant Women - Enhanced Usual Care Group (N=31) | Non-anxious Pregnant Women - Healthy Control (N=60)
Still birth (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 1 (1)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 12 (12) | 17 (17)
Child death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
The original sample size target was 300 for this biological supplement study. However, the study was delayed because of Covid-19 pandemic lockdowns in Pakistan and forced to end at the same time as the main study. This prevented us from collecting all the anticipated data, leaving us with a sample size of 117.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT04566861/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT04566861/ICF_001.pdf